CLINICAL TRIAL: NCT01640691
Title: A Clinical Study to Evaluate the Immunogenicity and Safety of Pandemic Influenza Vaccine, AdimFlu-W (H5N1), in Healthy Adults
Brief Title: Immunogenicity and Safety of Pandemic Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLUW001A
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Pandemic Influenza
Keywords: pandemic influenza; pandemic influenza vaccine; Influenza; Orthomyxoviruses; A/H5N1
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study vaccine (AdimFlu-W) (Experimental): 0.5 mL/dose, a total of 2 doses, 21 days apart
  Interventions: Biological: Pandemic Influenza Vaccine (H5N1)

INTERVENTIONS:
Biological: Pandemic Influenza Vaccine (H5N1) — Inactivated whole-virion vaccine
  1. Administration route: Intramuscular Injection
  2. Dosing schedule: 2 injections - at Day 1 and Day 22 separately
  3. Dose(s): Each dose (0.5 mL) contains the 15 mcg hemagglutinin (HA) of influenza A (A/Vietnam/1194/2004)
  Other Names: AdimFlu-W (H5N1) Pandemic Influenza Vaccine

SUMMARY:
The objectives of this single arm study are to evaluate the immune response and safety profiles of two injections of an inactivated whole-virion vaccine containing aluminum hydroxide adjuvant, AdimFlu-W (H5N1), against influenza A (H5N1) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant female (as indicated by a negative urine pregnancy test immediately on the day prior to first vaccine administration) between 20 to 60 years of age at the time of the first vaccination. Women of childbearing potential agree to practice highly effective birth control throughout the study (from Screening to Month 3).
* Subjects are free of obvious health problems as judged by investigator (established by medical history and physical examination) before entering the study.
* Subject is physically and mentally capable of participating in the study and willing to adhere to study procedures to complete all elements of the study diary.
* Subjects provide signed informed consent after receiving a detailed explanation of the study protocol prior to any study procedures.

Exclusion Criteria:

* Medical history of physician-confirmed infection with an H5N1 virus or a history of vaccination with an H5N1 influenza vaccine.
* Subject is at high risk of contracting H5N1 influenza infection (e.g. poultry workers).
* Has received any other licensed vaccines within 2 weeks for inactivated vaccines or 4 weeks for live vaccines prior to enrollment in this study.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Subject has used oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs within 30 days preceding the first dose of study vaccine.
* Subject has received a blood transfusion or immunoglobulins within 90 days prior to first dose of study vaccine, or planned administration of any blood products during the study period.
* Subject has a known allergy to eggs or other components of the study vaccine.
* Subject has a history of severe allergic reactions or anaphylaxis.
* Subject has a history of Guillain-Barré Syndrome.
* Subject has an acute illness or temperature greater than 38.0 degrees Celsius by any method within 3 days prior to each vaccination.
* Subject has confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Subject has a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating.
* Evidence of substance (alcohol or drug) abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Subjects with abnormal laboratory results at screening:(1) ALT or AST > or = 1 x upper limit of normal (ULN). (2) Creatinine > or = 1 x ULN. (3) Any significant laboratory abnormality as judged by the investigator
* Females are known pregnancy or a positive urine beta-human chorionic gonadotropin test result prior to the first study vaccine dose, or are lactating or nursing.
* Subject has any other condition that disqualifies his/her participation in the study in the opinion of the investigator.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2013-01-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Immunogenicity Endpoint: hemagglutination inhibition (HAI) titer and microneutralization (MN) titer | At Day 43 (21 days after the second dose).
  The primary immune response endpoint is to evaluate the seroconversion rate (SCR) in terms of HAI assays at Day 43 (21 days after the second dose).The secondary HAI endpoints are defined as following:
  1. SCR for the first vaccination, at Day 22.
  2. Seroprotection rates (SPR) for each vaccination, at Day 22 and 43.
  3. The geometric mean fold rise (GMFR) for each vaccination, at Day 22 and 43.
  The supportive immunogenicity endpoints of MN antibodies are SCRs, SPRs and GMFRs at Day 22 and 43.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events after vaccination. | At 4 weeks after two doses of study vaccine, 4 weeks apart. Reactogenicity will be recorded for 7 days after each vaccination.
  Safety data will consist of reactogenicity, serious and non-serious adverse events. Reactogenicity events are pre-specified adverse events systematically recorded for 7 days after each vaccination.The events included fever (≥38.0°C), runny nose or nasal congestion, cough, sore throat, muscle aches, headache, vomiting, nausea and malaise. Furthermore, the local (injection site) reactions were also evaluated, including soreness/pain, swelling, redness, ecchymosis and limitation of arm motion.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Jen Chang, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan